CLINICAL TRIAL: NCT06604728
Title: Evaluation of Effectiveness and Tolerance of Intravenous and Subcutaneous Biological Drugs in Gastrointestinal Diseases (BIOES)
Brief Title: Effectiveness and Tolerance of IV vs SC Biological Drugs in Gastrointestinal Diseases
Acronym: BIOES
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Scaldaferri Franco, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: BIOES - 5713
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients affected by IBD in therapy with biological therapies: cohort of patients affected by IBD in therapy with biological drugs, already subjected (retrospective cohort) or who will undergo (prospective cohort) for reasons of clinical practice to switch from the intravenous indication to the corresponding subcutaneous prescription (in particular, from vedolizumab or intravenous infliximab intravenously and to vedolizumab or subcutaneous infliximab).

SUMMARY:
Biologics are effective pharmacological treatments for Inflammatory Bowel Disease (IBD). To date, in the context of these pathologies, the formulations that can be administered subcutaneously are available for all the biological agents on the market (infliximab, adalimumab, golimumab, vedolizumab and ustekinumab) and can guarantee self-administration of the therapy at home with a reduction in hospital admissions , improved pharmacokinetics and pharmacoeconomic benefits For these reasons, the consolidation of the clinical practice of switching biological drugs to subcutaneous administration in patients with IBD in clinical remission could be a good strategy in terms of therapeutic efficacy and tolerability.

To date, intravenous and subcutaneous therapy for the biologics considered in the present study is considered equivalent both from a pharmacokinetic point of view ("bioequivalence" of the drug) and from a clinical point of view due to the available efficacy and safety data. The clinical choice of one or the other formulation generally takes into consideration the patient's concern, the subject's venous availability and the experience of the prescribing doctor. This protocol aims to collect the "real life" clinical experience and describe the clinical progress of the patients.

DETAILED DESCRIPTION:
The study is designed as a prospective, retrospective, 24-month observational cohort study. Patients' eligibility for enrolment will be assessed during the baseline visit at the Centre for Diseases of the Digestive System (CEMAD), Agostino Gemelli University Polyclinic Foundation IRCCS Università Cattolica del Sacro Cuore. Subjects meeting all inclusion criteria will be enrolled, and all subjects meeting at least one exclusion criterion will be excluded.

A cohort of patients suffering from IBD undergoing therapy with biological drugs, already undergoing (retrospective cohort) or who will undergo (prospective cohort) for clinical practice reasons a switch from the intravenous formulation to the corresponding subcutaneous formulation (in particular, from intravenous vedolizumab or infliximab to subcutaneous vedolizumab or infliximab) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Confirmed diagnosis of IBD (Crohn's disease, ulcerative colitis or indeterminate colitis)
* Intravenous therapy with vedolizumab or infliximab; OR
* Patients who for clinical reasons initiated subcutaneous vedolizumab or infliximab therapy at least 2 and up to 8 weeks after intravenous therapy with the same drugs for the prospective cohort and patients on subcutaneous vedolizumab and infliximab therapy for more than 8 weeks after intravenous therapy with the same drugs for the retrospective cohort;
* Stable (at least 12 weeks) steroid-free IBD clinical remission, defined as a finding of Harvey Bradshaw Index3 (HBI) scores < 5 or Partial Mayo Score 4.5 (PMS) < 2 for patients with Crohn's disease or colitis ulcerative, respectively, assessed at the time of switching the drug to subcutaneous administration;
* Ability to sign informed consent for participation in the study and to comply with the schedule of scheduled visits.

Exclusion Criteria:

* Patients with dietary or medication changes during the study period (for the prospective group) or who experienced dietary or medication changes in the 48 weeks between drug switching from intravenous to subcutaneous administration (for the retrospective group only) ;
* Patients undergoing colectomy or with cutaneous ostomy;
* Patients scheduled for hospitalization or surgery within the period of study participation;
* Concomitant enrollment in other interventional experimental protocols;
* Unstable personality or unable to adhere to protocol procedures;
* Any clinical condition which, in the opinion of the investigators, may contraindicate enrollment in the study;
* Refusal to sign informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who meet all the inclusion criteria, and all subjects who meet at least one exclusion criterion will be excluded. cohort of patients with IBD on biologic therapy, who have already undergone (retrospective cohort) or who will undergo (prospective cohort) for clinical practice reasons a switch from the intravenous formulation to the corresponding subcutaneous formulation (in particular, from vedolizumab or intravenous infliximab intravenously and to vedolizumab or subcutaneous infliximab).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who maintain clinical remission | 24 months
  percentage of patients who maintain clinical remission after switching to subcutaneous therapy without further changes in current therapy

CONTACTS AND LOCATIONS:
Overall Officials: Franco Scaldaferri, PI, Principal Investigator — Fondazione Policlinico Gemelli, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC CEMAD, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided